CLINICAL TRIAL: NCT04126096
Title: The Negative Predictive Value and Non-irritant Skin Testing Concentrations of Beta-Lactam Containing Antibiotics Other Than Penicillin.
Brief Title: Negative Predictive Value and NIC of Beta-Lactam Antibiotics.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Alexei Gonzalez-Estrada, MD, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-002587
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Skin testing
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Group (Experimental): Study team is developing a new diagnostic skin testing procedure for patients who receive beta lactam containing antibiotics during surgery (other than penicillin) in order to determine Negative Predictive Values and Non-Irritant Concentrations.
  Interventions: Diagnostic Test: Skin Testing beta-lactams

INTERVENTIONS:
Diagnostic Test: Skin Testing beta-lactams — Percutaneous skin prick followed by Intradermal Injections of NMBAs at increasing concentrations compared with an established positive and negative control.

SUMMARY:
The researchers are trying to evaluate how much medication is required for allergy skin testing and to determine the likelihood that patients with a negative test truly don't have an allergy to the tested drug of skin testing to commonly used antibiotics.

DETAILED DESCRIPTION:
This study will be a prospective study to accurately determine the negative predictive value of skin testing with beta lactam containing antibiotics other than penicillin .

It is hypothesized that the concentrations that should be used for beta lactams are actually much lower than previously recommended and that the higher incidence of identifiable beta lactam induced allergic reactions during anesthesia in the past may be due to irritation of the skin rather than a true allergic reaction (false positives).

ELIGIBILITY:
Inclusion Criteria:

* All adults > or = to 18 y/o undergoing surgery

Exclusion Criteria:

* Minors under the age of 18 y/o, Adults unable to consent, or those Adults with previous allergic reaction history during previous surgeries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 747 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Non-Irritant Concentrations to common beta lactam containing antibiotics other than penicillin | 1 Year
  Determine the NIC to common beta lactam containing antibiotics

SECONDARY OUTCOMES:
Negative Predictive Value of Intradermal Skin Testing to commonly used beta lactam containing antibiotics other than penicillin | 1 Year
  Determine Negative Predictive Value of Intradermal Skin Testing to commonly used beta lactam containing antibiotics

OTHER OUTCOMES:
Max Concentration used when skin testing to beta lactam containing antibiotics other than penicillin | 1 Year
  Close gap on the variability of the maximal concentration used when skin testing beta lactam containing antibiotics.

CONTACTS AND LOCATIONS:
Overall Officials: Alexei Gonzalez Estrada, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials